CLINICAL TRIAL: NCT01116869
Title: A Multi-Center, Prospective Study to Evaluate the Ability of CTC Enumeration Using the CellSearch® Circulating Tumor Cell Kit to Predict Prognosis and to Assess the Agreement Between CTC and Imaging Determined Response in MBC Patients 一项评价CellSearch® 循环肿瘤细胞检测试剂盒对复发转移性乳腺癌患者进行循环肿瘤细胞检测 以预测病人预后的能力及循环肿瘤细胞检测和影像学疗效判断之间一致性的多中心、前瞻性的研究
Brief Title: China CellSearch Study
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Medical, China (Industry)
Responsible Party: Sponsor
Other Study IDs: 200901
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Breast Cancer; Benign Breast Disease
Keywords: MBC; Healthy; Benign disease; Confirmed metastatic breast cancer patient with at least one measurable solid tumor according to the RECIST guideline; Medical examinations detect no breast benign and malignant tumors; Benign Breast Disease; Pathology diagnosed breast benign tumor disease
MeSH Terms: conditions — Breast Neoplasms; Cystic Fibrosis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- MBC patients: 300 MBC patients, each of whom will provide a series of at least 3 blood draws (baseline, 3-4 weeks and 6-8 weeks after the initiation of the systemic therapy) for CTC analysis, will be enrolled. All MBC patients will be followed for a maximum of 36 months for disease progression and survival.
- Benign disease volunteers: 100 Benign disease volunteers whom will donate blood 1 time for CTC analysis, will be enrolled as controls.
- Healthy volunteers: 100 Healthy volunteers whom will donate blood 1 time for CTC analysis, will be enrolled as controls.

SUMMARY:
The study is designed to confirm the current indication (below) of the CellSearch® Circulating Tumor Cell Kit in metastatic breast cancer (MBC) patients for use of the kit in China.

The CellSearch® Circulating Tumor Cell Kit is intended for the enumeration of circulating tumor cells (CTC) of epithelial origin (CD45-, EpCAM+, and cytokeratins 8, 18+, and/or 19+) in whole blood.

The presence of CTC in the peripheral blood, as detected by the CellSearch® Circulating Tumor Cell Kit, is associated with decreased progression free survival and decreased overall survival in patients treated for metastatic breast cancer. This test is to be used as an aid in the monitoring of patients with metastatic breast cancer. Serial testing for CTC should be used in conjunction with other clinical methods for monitoring metastatic breast cancer. Evaluation of CTC at any time during the course of disease allows assessment of patient prognosis and is predictive of progression free survival and overall survival.

DETAILED DESCRIPTION:
A longitudinal, multi-center, prospective study will be conducted in MBC patients to evaluate the ability of CTC to predict the patients' prognosis. A separate population of healthy and benign disease subjects will serve as controls to compare the CTC incidence in this control group versus the MBC group at baseline. Correlation between CTC and radiographic response to the systemic therapies in the MBC study group will also be assessed.

300 MBC patients, each of whom will provide a series of at least 3 blood draws (baseline, 3-4 weeks and 6-8 weeks after the initiation of the systemic therapy) for CTC analysis, will be enrolled. All MBC patients will be followed for a maximum of 36 months for disease progression and survival.

200 healthy and benign disease volunteers, each of whom will donate blood 1 time for CTC analysis, will be enrolled as controls.

ELIGIBILITY:
Inclusion Criteria

* Female
* over 18 and less than 70 years of age
* Subject having agreed to participate in the study and follow the study procedures by providing written informed consent prior entering the study.
* For MBC Subject Set only Confirmed metastatic breast cancer patient with at least one measurable solid tumor according to the RECIST guideline Starting a new line of systemic therapy which is recommended in the Chinese edition of NCCN Clinical Practice Guidelines in Oncology Breast Cancer Guideline 2009 line of chemotherapy should be over 3 ECOG performance grade of 0 to 2 Life expectancy over 3 months
* For Healthy Subject Set only Medical examinations detect no breast benign and malignant tumors
* For Benign Breast Disease Subject Set only Pathology diagnosed breast benign tumor disease

Exclusion Criteria

* Self reported pregnancy
* For MBC Subject Set only Prior history of other malignancy Patients who have surgery to remove any metastatic lesions or receive radiation therapy during her participation in the study
* For Healthy Subject Set only Prior history of breast benign tumor disease or any malignancy Any conditions inappropriate for blood drawing
* For Benign Breast Disease Subject Set only Prior history of any malignancy Any conditions inappropriate for blood drawing

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The hazard ratio of disease progression in patients with unfavorable versus favorable CTC counts at baseline, 3-4 weeks and 6-8 weeks after the initiation of therapy will be estimated using Cox regression.
  Kaplan-Meier plots for PFS will be constructed using the favorable and unfavorable CTC patient groups. The log-rank test will be used to determine if the curves for the two CTC groups are statistically significantly different.
  The hazard ratio of death in patients with unfavorable versus favorable CTC counts at each blood draw time point will be estimated using Cox regression. Kaplan-Meier plots for OS will be constructed using the favorable and unfavorable CTC patient groups.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-03-25 (Actual); Primary Completion 2011-06-22 (Actual); Study Completion 2014-01-06 (Actual)

PRIMARY OUTCOMES:
Ability of CTC levels to predict progression-free survival (PFS) in MBC patients. | 12 months

SECONDARY OUTCOMES:
Ability of CTC levels to predict overall survival (OS) in MBC patients. | 3 years
Agreement between CTC counts (3-4 weeks and 6-8 weeks) after the initiation of a new line of systemic therapy and the patient's response as determined by imaging evaluation (6-8 weeks after the initiation of therapy) in MBC patients. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, Doctor, Study Chair — 307 Hosptial of PLA; Zhimin Shao, Doctor, Principal Investigator — Shanghai Cancer Hosptial; Tao Ouyang, Doctor, Principal Investigator — Beijing Cancer Hosptial; Erwei Song, Doctor, Principal Investigator — Zhongshan 2nd Hospital; Ning Liao, Doctor, Principal Investigator — The Second People's Hospital of GuangDong Province; Xiaojia Wang, Doctor, Principal Investigator — Zhejiang Cancer Hosptial; Zhongsheng Tong, Doctor, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- 307 Hosptial of PLA, Beijing, China